CLINICAL TRIAL: NCT05279924
Title: Impact of Implementation of Prophylaxis With Emicizumab in Children With Severe Hemophilia A in Ivory Coast
Brief Title: Outcomes of Prophylaxis With Emicizumab in Children With Severe Hemophilia A in Ivory Coast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Lambert Catherine, Clinical Professor. Hematology department, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001-22/MSHPCMU/CNESVS-km
Record Dates: First submitted 2022-02-25; First posted 2022-03-15 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Intervention Model Description: outcomes of prophylaxis with Emicizumab in Ivoirian boys with severe hemophilia A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivoirian Boys with severe Hemophilia A treated with Emicizumab (Experimental): All Ivoirian boys with severe Hemophilia A (with and without inhibitors) on prophylaxis with Emicizumab
  Interventions: Drug: Prophylaxis with Emicizumab

INTERVENTIONS:
Drug: Prophylaxis with Emicizumab — Prophylaxis with Emicizumab in Ivoirian boys with severe hemophilia A

SUMMARY:
Assessment of the outcomes of prophylaxis with Emicizumab in children with severe hemophilia A in Ivory Coast

DETAILED DESCRIPTION:
Assessment of the outcomes of prophylaxis with Emicizumab in children with severe hemophilia A in Ivory Coast.

Duration of the study: 1 year after initiation of prophylaxis with Emicizumab

Inclusion criteria: boys aged > 2 years, affected with severe hemophilia A with or without inhibitors

Evaluated outcomes: annual bleeding rate, days of absence from school, the need for additional facteur VIII consumption, satisfaction about the treatment and quality of life.

Tools used to assess quality of life are the Ivoirian version of the Canadian Haemophilia Outcomes-Kids' Life Assessment Tool version 2 (CHO-KLAT) and EQ-5D

The satisfaction of the parents will be assessed using the patients' global impression of change scale (PGIC).

ELIGIBILITY:
Inclusion Criteria: severe hemophilia A with or without inhibitors -

Exclusion Criteria: parents refusal

-

Ages: 2 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Change in annual bleeding rate | change in annual bleeding rate from baseline at 6 months and 12 months
  Using the patients' logbook
Change in the scores of HR-QoL tools CHO-KLAT and EQ-5D in children treated with Emicizumab | Change in the scores of HR-QoL tools CHO-KLAT and EQ-5D at 6 months.
  Using the CHO-KLAT and EQ-5D. The scales range from 0 to 100 with 0 representing the worst quality of life and 100 the best quality of life score
Satisfaction of the parents about the treatment with Emicizumab after 6 month | Assessment at 6 months after initiation of Emicizumab
  Usign the PGIC (scale ranging from extremely satisfied to extremely unsatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: N'Dogomo Meité, MD, Principal Investigator — CHU de Cocody
Locations (1):
- CHU de Yopougon, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: No